CLINICAL TRIAL: NCT02948504
Title: Treatment of Small Unruptured Intracranial Aneurysms Based on Clinical Characteristics, Morphology and Hemodynamic Features
Brief Title: Chinese Small Intracranial Aneurysm Study (CSIAS)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RJ2016144K1.0
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Intracranial Aneurysm; Unruptured Cerebral Aneurysm; Treatment Side Effects
Keywords: Unruptured Intracranial Aneurysm; Small aneurysms; Risk of rupture; Natural history; Endovascular Coiling; Surgical clipping
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Observation: Aneurysms are left untreated based on patients and family's wishes. These patients will be included in the observation group.
- Coiling or Clipping: Patients are included in the coiling group if they undergo endovascular coiling, such as single coiling, stent-assisted coiling and balloon-assisted coiling. Or Patients are included in the clipping group if they undergo surgical coiling, such as aneurysm neck clipping, aneurysm isolation or trapping.
  Interventions: Procedure: Coiling or Clipping

INTERVENTIONS:
Procedure: Coiling or Clipping — All patients are treated under general anesthesia and systemic heparinization. A bolus of 50-75 IU/kg of heparin is given after femoral sheath placement, and intermittent boluses of 1250 IU per hour are given during the procedure. Activated clotting time is maintained at 2-3 times baseline level. Balloon-assisted coiling or stent-assisted coiling are considered in aneurysms with an unfavorable morphology (aneurysm neck≥ 4.0 mm or dome/neck ≤2.0). All anterior circulation aneurysms are clipped through a standard pterional or frontal temporal approach. The posterior circulation aneurysms are treated using far lateral approach depending on the aneurysm location.
  Groups: Coiling or Clipping

SUMMARY:
Intracranial aneurysms are common in the general population. The overall prevalence of unruptured intracranial aneurysms (UIAs) is estimated of 2.3-3.2% in the population without specific risk factors for SAH. As noninvasive imaging modalities are more commonly used than before, UIAs are increasingly being detected. Most patients with small aneurysms (less than 5mm) are incidentally found in clinical practice. Some studies indicate that the majority of patients with UIAs, particularly with small aneurysms (<7mm), have a low risk of rupture, and others have found that small ruptured aneurysms have a high proportion in patients with SAH. Therefore, there is a lot of controversy regarding which small aneurysms can be left untreated, or which aneurysms are needed to be treated with clipping or coiling.

The prevalence varies widely among different detection methods, race/ethnicity or patients with other inherited diseases. Although a wealth of data is available for the natural history of UIAs, the true natural history remains unknown because case selection bias occur in almost all studies. However, data on Chinese UIA is unknown. Using the MR angiography (MRA) to detect aneurysms, the prevalence is 7% of selected adult population in China. Therefore, small UIAs are very common and are increasingly being detected in clinical practice. Conservative treatment, surgical clipping and endovascular coiling are the three treatment options for UIAs. The optimal treatment remains controversial, particularly for small aneurysms (less than 7mm). To date, no clinical trials have compared the safety and efficacy between conservative treatment and surgical clipping or endovascular coiling for UIAs. It may be impossible to conduct the randomized controlled study considering aneurysm ruptured as a devastating event. However, surgical clipping or endovascular treatment itself carries a risk of immediate morbidity or mortality. Therefore, a substantial variability widely exists in treatment decision-making for UIAs, and this may lead to a great variability in clinical recommendations.

Our study is a prospective observational study to identify the incidence of rupture of small aneurysms in the first year after the diagnosis of the aneurysm which is left untreated. Meanwhile, we determine the differences of outcomes, procedural complications, and rates of retreatment between surgical clipping and endovascular coiling for small UIAs in China.

DETAILED DESCRIPTION:
1. Background: There is a lot of controversy regarding which aneurysms can be left untreated, or which aneurysms are needed to be treated with clipping or coiling. To date, no clinical trials have compared the safety and efficacy between conservative treatment and surgical clipping or endovascular coiling for small UIAs.
2. Study design: A multicenter prospective observation registry study. This study is undertaken to conform to the study protocol. Patients will be recruited between December 2016 and December 2018. Patients are eligible for the study if they meet the inclusion criteria and they are not eligible if any of the following exclusion criteria are met.
3. Procedures: All patients were interviewed by a multidisciplinary team that consisted of vascular neurosurgeons, interventional neuroradiologists and anesthetists. If patients meet all of the inclusion criteria: an unruptured aneurysms ≤5mm are enrolled and then followed up at 6 and12 months. Clinical observation, surgical clipping and endovascular coiling are the three treatment options for UIAs. In general, when an UIA is detected, it should be needed to quit smoking, to aggressively manage hypertension, and to control alcohol use. When an aggressive treatment is considered, treatment risks should be balanced against the risk of rupture.

ELIGIBILITY:
Inclusion Criteria:

1. Intracranial unruptured aneurysms confirmed by digital subtraction angiography DSA, CT angiography or MR angiography (MRA);
2. The maximum size of unruptured aneurysm ≤5mm;
3. Informed consent

Exclusion Criteria:

1.Patients with severe systemic disorders and expected life span less than one year; 2.Pregnant or lactating women.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Five hundred patients with unruptured aneurysms will registered in this study during the 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Rupture of an unruptured aneurysm | One year of follow-up
  These aneurysms are left untreated.

SECONDARY OUTCOMES:
Regrowth of an unruptured aneurysm | 9 and 12 months of imaging follow-up
Recurrence and retreatment after coiling or clipping | one year of follow-up
Poor outcome after coiling or clipping | 6 and 12 months
  Poor outcome is defined as a mRS 3-6

OTHER OUTCOMES:
Procedural complications | 30 days after coiling or clipping

CONTACTS AND LOCATIONS:
Overall Officials: Jieqing Wan, MD,PHD, Principal Investigator — Department of Neurosurgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sonobe M, Yamazaki T, Yonekura M, Kikuchi H. Small unruptured intracranial aneurysm verification study: SUAVe study, Japan. Stroke. 2010 Sep;41(9):1969-77. doi: 10.1161/STROKEAHA.110.585059. Epub 2010 Jul 29. PMID 20671254
- [Background] Rahman M, Smietana J, Hauck E, Hoh B, Hopkins N, Siddiqui A, Levy EI, Meng H, Mocco J. Size ratio correlates with intracranial aneurysm rupture status: a prospective study. Stroke. 2010 May;41(5):916-20. doi: 10.1161/STROKEAHA.109.574244. Epub 2010 Apr 8. PMID 20378866
- [Background] Greving JP, Wermer MJ, Brown RD Jr, Morita A, Juvela S, Yonekura M, Ishibashi T, Torner JC, Nakayama T, Rinkel GJ, Algra A. Development of the PHASES score for prediction of risk of rupture of intracranial aneurysms: a pooled analysis of six prospective cohort studies. Lancet Neurol. 2014 Jan;13(1):59-66. doi: 10.1016/S1474-4422(13)70263-1. Epub 2013 Nov 27. PMID 24290159
- [Background] Brown RD Jr, Broderick JP. Unruptured intracranial aneurysms: epidemiology, natural history, management options, and familial screening. Lancet Neurol. 2014 Apr;13(4):393-404. doi: 10.1016/S1474-4422(14)70015-8. PMID 24646873
- [Background] Juvela S, Poussa K, Lehto H, Porras M. Natural history of unruptured intracranial aneurysms: a long-term follow-up study. Stroke. 2013 Sep;44(9):2414-21. doi: 10.1161/STROKEAHA.113.001838. Epub 2013 Jul 18. PMID 23868274
- [Background] Guresir E, Vatter H, Schuss P, Platz J, Konczalla J, de Rochement Rdu M, Berkefeld J, Seifert V. Natural history of small unruptured anterior circulation aneurysms: a prospective cohort study. Stroke. 2013 Nov;44(11):3027-31. doi: 10.1161/STROKEAHA.113.001107. Epub 2013 Sep 3. PMID 24003049
- [Background] UCAS Japan Investigators; Morita A, Kirino T, Hashi K, Aoki N, Fukuhara S, Hashimoto N, Nakayama T, Sakai M, Teramoto A, Tominari S, Yoshimoto T. The natural course of unruptured cerebral aneurysms in a Japanese cohort. N Engl J Med. 2012 Jun 28;366(26):2474-82. doi: 10.1056/NEJMoa1113260. PMID 22738097
- [Background] Tominari S, Morita A, Ishibashi T, Yamazaki T, Takao H, Murayama Y, Sonobe M, Yonekura M, Saito N, Shiokawa Y, Date I, Tominaga T, Nozaki K, Houkin K, Miyamoto S, Kirino T, Hashi K, Nakayama T; Unruptured Cerebral Aneurysm Study Japan Investigators. Prediction model for 3-year rupture risk of unruptured cerebral aneurysms in Japanese patients. Ann Neurol. 2015 Jun;77(6):1050-9. doi: 10.1002/ana.24400. Epub 2015 Apr 22. PMID 25753954
- [Background] Murayama Y, Takao H, Ishibashi T, Saguchi T, Ebara M, Yuki I, Arakawa H, Irie K, Urashima M, Molyneux AJ. Risk Analysis of Unruptured Intracranial Aneurysms: Prospective 10-Year Cohort Study. Stroke. 2016 Feb;47(2):365-71. doi: 10.1161/STROKEAHA.115.010698. Epub 2016 Jan 7. PMID 26742803